CLINICAL TRIAL: NCT05926219
Title: Skeletal Muscle Myosin Binding Protein C in Fatigue and Aging
Brief Title: C-Protein in Fatigue and Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: Wu Tsai Human Performance Alliance (Unknown); National Institutes of Health (NIH) (NIH); Oregon Health and Science University (Other); Washington State University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11262017.042; R21AG077125-01 (NIH)
Record Dates: First submitted 2023-05-31; First posted 2023-07-03 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-01

CONDITIONS: Aging; Muscle Atrophy or Weakness; Sarcopenia in Elderly; Sarcopenia
Keywords: muscle; aging; elderly; myosin; protein; sarcomere; exercise; function; atrophy; contractile; strength; balance; mobility; MyBP-C; fiber; biopsy; skeletal muscle; fatigue
MeSH Terms: conditions — Muscular Atrophy; Asthenia; Sarcopenia; Motor Activity; Atrophy; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fatigue (Experimental): Volunteers will perform one-legged knee extension exercise until fatigue while seated on an ergometer. Volunteers will then undergo bilateral skeletal muscle biopsies of the vastus lateralis muscle in their thigh.
  Interventions: Behavioral: Fatiguing Exercise

INTERVENTIONS:
Behavioral: Fatiguing Exercise — Volunteers will perform knee extension exercise of the dominant limb while seated in a chair designed for exercise of the knee extensor muscle group. The chair will be equipped with a lever arm, aligned with the axis of rotation of the knee and fixed to the distal shank, 2 centimeters proximal to the ankle joint. The lever arm will be instrumented to provide resistance and measure velocity. The volunteers will perform 3-5 maximum voluntary contractions (MVC) to determine peak torque. Once established, volunteers will rest for 5 minutes before initiating the fatigue protocol, whereby they will perform repeated MVC of the dominant limb against resistance equal to or less than 50% of MVC until range of motion cannot be maintained. Because the goal of this exercise is to uniformly fatigue the quadriceps muscle group, this exercise will be performed continuously. It is expected to take between 1 and 3 minutes to achieve the desired level of fatigue.

SUMMARY:
This study is investigating changes to the proteins in skeletal muscle that contribute to reduced muscle size and muscle function that occurs with aging.

DETAILED DESCRIPTION:
Age-related muscle atrophy and contractile dysfunction have been well described at the cellular level, but the molecular mechanisms that contribute to this dysfunction are poorly understood. Improved understanding of these mechanisms is critically important for the improvement of physical rehabilitation in older adults at risk for mobility impairment and physical disability. Our studies will pursue pre-clinical evidence that post translational modification of specific proteins in skeletal muscle lead to an "aging phenotype" in skeletal muscle that may unlock new strategies for improving physical function in older adults with physical frailty.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages 18-35 or 65-80 years
* Healthy by self-report
* Willing to participate in all aspects of the study design including muscle biopsy, unilateral exercise, and physical activity monitoring
* Fluent in English (due to lack of translation services, it is not practical to conduct the study using a language other than English).

Exclusion Criteria:

* Orthopaedic limitation (severe knee osteoarthritis, prior joint replacement, etc.).
* Volunteer has dementia or related mental issues that potentially put the subject at risk as determined by prior diagnosis.
* Volunteer has known untreated endocrine disease (hypo/hyper thyroidism, Addison's Disease or Cushing's syndrome, etc.)
* Volunteer has untreated/poorly-controlled hypertension (stage 2, per American College of Cardiology [>140/90 mmHg]).
* Volunteer has significant heart, liver, kidney or respiratory disease.
* Volunteer has diabetes (insulin dependent or non-insulin dependent).
* Volunteer has known coagulopathies.
* Volunteer has taken anabolic steroids in the prior six months.
* Volunteer has received treatment for cancer (other than effective Mohs Surgery for successful removal of basal cell or squamous cell carcinomas)
* Unexpected weight loss >5kg is last 12 months
* Volunteer is an active smoker or quit within the last year.
* Volunteer has known current alcohol or drug use disorder (AUD; defined as binge drinking of >4 days in the last month. Binge drinking is >5 drinks for men and >4 drinks for women, per occasion). Or, if a volunteer reports drinking in excess of "low risk" per NIAAA (>7 drinks/week for men and >3 drinks/day for women and >14 drinks/week and >4 drinks/day).
* Volunteer has a diagnosed neuromuscular disorder.
* Volunteer has allergy to lidocaine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Phosphorylation of myosin binding protein c (MyBP-C) | One week after the participant undergoes the biopsies.
  Muscle tissue is immediately frozen after biopsy. Liquid chromatography and high resolution mass spectrometry will be used to do a full analysis of the phosphorylation sites on MyBP-C isolated from the biopsied muscle tissue.

SECONDARY OUTCOMES:
Muscle fiber Force | Within three weeks of the intervention and biopsies.
  Ex vivo assessment of Force (mN) will be performed on muscle fibers and bundles isolated from fatigued and non-fatigued muscle biopsies.
Muscle fiber Tension | Within three weeks of the intervention and biopsies.
  Ex vivo assessment of Tension (kPa) will be performed on muscle fibers and bundles isolated from fatigued and non-fatigued muscle biopsies.
Muscle fiber Velocity | Within three weeks of the intervention and biopsies.
  Ex vivo assessment of Velocity (Lo/s) will be performed on muscle fibers and bundles isolated from fatigued and non-fatigued muscle biopsies.
Muscle fiber Power | Within three weeks of the intervention and biopsies.
  Ex vivo assessment of Power (w/L) will be performed on muscle fibers and bundles isolated from fatigued and non-fatigued muscle biopsies.

CONTACTS AND LOCATIONS:
Overall Officials: Damien M Callahan, Ph.D., Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT05926219/Prot_ICF_000.pdf